CLINICAL TRIAL: NCT02346279
Title: Study to Evaluate the Responsiveness and Minimal Clinical Important Difference (MCID) of the 'Multiple Sclerosis Questionnaire for Physiotherapists' (MSQPT)
Brief Title: Responsiveness and Minimal Clinical Important Difference of the Multiple Sclerosis Questionnaire for Physiotherapists
Status: Completed | Type: Observational
Sponsor: Institut fuer Physiotherapieforschung (Other)
Collaborators: Schweizer Physiotherapie Verband physioswiss (Unknown); Schweizerische Multiple Sklerose Gesellschaft (Other)
Responsible Party: Sponsor
Other Study IDs: Responsivität und MCID MSQPT
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Rehabilitation; Questionnaire; Patient-Reported Outcome; Responsiveness; Minimal Important Clinical Difference
MeSH Terms: conditions — Multiple Sclerosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Persons in physical therapy treatment: Questionnaires (MSQPT, HAQUAMS, Transition Questionnaire for Patient and treating physiotherapist), physical tests (9HPT, 6MTWT, BBS, 6MWT), EDSS
  Interventions: Other: Questionnaires, EDSS, physical test

INTERVENTIONS:
Other: Questionnaires, EDSS, physical test — 6 Meter timed walking test, Nine Hole Peg Test, Berg balance Scale, MSQPT, HAQUAMS, Transition Questionnaire for Patients, Transition Questionnaire for Therapists, EDSS, 6 Minute Walking Test

SUMMARY:
The aim of this survey is the evaluation of the responsiveness and the estimation of the MCID of the German and French Multiple Sclerosis Questionnaire for Physiotherapists, a self-rating Patient Reported Outcome questionnaire. This multicenter project uses a combined anchor and distribution based approach with multiple anchors to provide a range of MCID estimates or a single MCID for the reliable and valid Items, Activity and Participation group and the Total Score of the MSQPT, which should to be used as guidelines in daily practice.

DETAILED DESCRIPTION:
The MSQPT is a highly reliable and valid questionnaire that was designed to be an aid for physiotherapists to asses the course of treatment of Persons with MS (PwMS). The assessment of the responsiveness of the MSQPT, which is so crucial for the evaluative value of an instrument used in long time treatment of PwMS, is the focus of this study.

This multicenter study uses a convenience sample of 81 PwMS, who are in short or long term treatment widespread over Switzerland. At baseline, the testers record age, gender, type of MS and disease duration since diagnosis. The tests will be executed in the following order: six-meter Timed Walking Test (6MTWT), nine-hole peg test (9HPT), Berg Balance Scale (BBS), MSQPT, Hamburg Quality of Life Questionnaire in Multiple Sclerosis (HAQUAMS), Expanded Disability Status Scale (EDSS) and Transition Questionnaires for the Patient and the treating physiotherapist. Finally the six-minute walk (6MWT) rest will be carried out. The intervention with long term patients was planned every next 6 months after the baseline testing (T1, T2 and T3). The short time patient will be tested at base line and after 3 to 4 months or at the end of the rehabilitation period (T1).

A standardized test protocol manual will be used by the experienced and trained testers.

Effect Size , Standardized Response Mean (SRM). Modified SRM (MSRM), Relative Efficiency (RE), Sensitivity and Specificity and correlation estimates will describe the anchor based responsiveness. The combined anchor and distribution based approach is used in search of a MCID. The distribution based approach uses statistics like Standard Deviation, Standard Error of Measurement and Minimal Detectable Change as indicators of MCID. The anchor based approach uses global ratings of change out of the perspective of the patient and the physiotherapist for different aspects of health: general health status, balance, walking ability, arm function, fatigue, pain, amount of being active, participation in social life and general impairment due to MS. Minimal change is defined as one to two gradient change on the 9 point scale of the transition questions. The expected wide range of MCIDs will be narrowed to a small range or single MCID by triangulation and selection of the MCID with best selectivity and specificity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosed MS, who are in physiotherapeutic treatment because of MS, older than 18 year, must be able to read the MSQPT by himself, native language German or French, EDSS score of less or equal 6.5

Exclusion Criteria:

* Acute episode of MS, grave cognitive changes, bedfast patient, distinct fatigue, able to perform less than 2 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons suffering from Multiple Sclerosis that are in physical therapy treatment because of the multiple sclerosis and are treated in private practice or in ambulant department of hospitals in the German part of Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2011-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Multiple Sclerosis Questionnaire for Physical Therapists | 20 minutes
  Items 'Taking a Shower', 'Getting in and out of a car', 'Walking distance' and Walking Time', Activity Group, Participation Group, Total Sum of Items

SECONDARY OUTCOMES:
6 Meter Timed Walking Test | 3 to 20 seconds
  Walking 6 Meter, static start, walking at normal speed with or without an walking aid, average of three repetitions
Nine Hole Peg Test | up to 5 minutes
  Putting as fast as possible nine pegs, one after the other, in nine holes and put them back, one after the other, in the container, best of 2 repetitions
Berg Balance Scale | 20 minutes
  14 Standardized tests, the Gold standard in Balance testing
Hamburg Quality of Life Questionnaire in Multiple Sclerosis | 20 minutes
  Patient Reported Quality of Life Questionnaire
Expanded Disability Status Scale | 5 minutes
  Gold standard in describing the status of MS
6 Minutes Walking Test | 6 minutes
  Walking 6 minutes as far the person can walk, static start, walking at normal speed with or without walking aid

CONTACTS AND LOCATIONS:
Overall Officials: Nanco van der Maas, Principal Investigator — Institut für Physiotherapieforschung

REFERENCES:
- [Background] Fitzpatrick R, Davey C, Buxton MJ, Jones DR. Evaluating patient-based outcome measures for use in clinical trials. Health Technol Assess. 1998;2(14):i-iv, 1-74. No abstract available. PMID 9812244
- [Background] Gold SM, Heesen C, Schulz H, Guder U, Monch A, Gbadamosi J, Buhmann C, Schulz KH. Disease specific quality of life instruments in multiple sclerosis: validation of the Hamburg Quality of Life Questionnaire in Multiple Sclerosis (HAQUAMS). Mult Scler. 2001 Apr;7(2):119-30. doi: 10.1177/135245850100700208. PMID 11424632
- [Background] Learmonth YC, Paul L, McFadyen AK, Mattison P, Miller L. Reliability and clinical significance of mobility and balance assessments in multiple sclerosis. Int J Rehabil Res. 2012 Mar;35(1):69-74. doi: 10.1097/MRR.0b013e328350b65f. PMID 22315143
- [Background] Revicki D, Hays RD, Cella D, Sloan J. Recommended methods for determining responsiveness and minimally important differences for patient-reported outcomes. J Clin Epidemiol. 2008 Feb;61(2):102-9. doi: 10.1016/j.jclinepi.2007.03.012. Epub 2007 Aug 3. PMID 18177782
- [Background] Wyrwich KW, Norquist JM, Lenderking WR, Acaster S; Industry Advisory Committee of International Society for Quality of Life Research (ISOQOL). Methods for interpreting change over time in patient-reported outcome measures. Qual Life Res. 2013 Apr;22(3):475-83. doi: 10.1007/s11136-012-0175-x. Epub 2012 Apr 17. PMID 22528240
- [Derived] van der Maas NA. Patient-reported questionnaires in MS rehabilitation: responsiveness and minimal important difference of the multiple sclerosis questionnaire for physiotherapists (MSQPT). BMC Neurol. 2017 Mar 16;17(1):50. doi: 10.1186/s12883-017-0834-1. PMID 28302081